CLINICAL TRIAL: NCT05857774
Title: Respiratory Muscle Structure and Function in Mechanically Ventilated Patients and Long-term Outcomes
Acronym: RESPIRE
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5875
Record Dates: First submitted 2023-03-02; First posted 2023-05-15 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Mechanical Ventilation Complication; Diaphragm Injury; Lung Injury; Respiratory Insufficiency; Abdominal Muscle Strained
MeSH Terms: conditions — Lung Injury; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skeletal Troponin-I
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases: Adult patients ≥18 years of age undergoing invasive mechanical ventilation in the ICU for any reason within 36 hours of intubation
  Interventions: Other: Sonographic measurements; Other: Physiological measurements; Other: Biological measurements
- Control condition A: Non-invasively ventilated patients in the ICU within 36 hours of initiating non-invasive ventilation
  Interventions: Other: Sonographic measurements; Other: Physiological measurements; Other: Biological measurements
- Control condition B: Non-ventilated patients admitted to the ICU receiving no respiratory support or oxygen therapy alone, including high flow nasal cannula
  Interventions: Other: Sonographic measurements; Other: Physiological measurements; Other: Biological measurements

INTERVENTIONS:
Other: Sonographic measurements — Diaphragm thickness, diaphragm tidal thickening fraction, abdominal muscle thickness, rectus femoris cross-sectional area, maximal diaphragm thickening fraction, abdominal muscle thickening fraction
Other: Physiological measurements — Airway occlusion pressure, maximal inspiratory pressure, muscle research council score
Other: Biological measurements — Skeletal troponin-I

SUMMARY:
Air is normally pumped in and out of the lungs by the muscles that contribute to inhalation and exhalation, called the respiratory muscles. The abdominal muscles help by forcing air out of your lungs during exhalation; whereas the diaphragm, the main muscle used for breathing, contracts to get air into the lungs during inhalation. With mechanical ventilation, respiratory muscles are able to rest and recover while the breathing machine takes over; however, this may cause respiratory muscle weakness. Patients who develop weakness of these muscles may require more assistance from the ventilator and take longer to recover their ability to breathe without assistance. The impact of this phenomenon on long-term outcomes is uncertain.

The RESPIRE study is designed to characterize how respiratory muscles change during mechanical ventilation and to evaluate the impact on long term quality of life. An additional objective of this study is to examine novel measures obtained from automated functions of a ventilator, that may better predict success from weaning from mechanical ventilation.

DETAILED DESCRIPTION:
Previous work has established that diaphragm atrophy during mechanical ventilation is associated with adverse clinical outcomes. Abdominal muscles, which are engaged during breathing also undergo atrophy during mechanical ventilation. However, the relationship between these muscles and how they relate to long term function status is known and warrants further investigation.

Mechanical ventilation is a life-saving technique in patients with respiratory failure, however reasons why some patients require long term ventilation and are unsuccessful from weaning from ventilators are not fully elucidated. Respiratory muscle dysfunction as a result of mechanical ventilation is only recently being understood. Diaphragm atrophy is associated with adverse clinical outcomes, but the same is unknown if this holds true with abdominal muscle atrophy. Properly understanding the natural progression of diaphragm and abdominal muscle atrophy and dysfunction, and how they relate to each other, is critical to identifying markers or factors that may put particular patients at risk for long durations of mechanical ventilation and adverse clinical outcomes.

This study will provide important insights into the relationship between inspiratory and expiratory muscle function, and the evolution of functional impairments in critical care patients undergoing weaning from invasive mechanical ventilation. Further understanding of the pathophysiological processes of how these muscle groups interact in this context is important in moving forward with potential therapeutic strategies aimed at mitigating injury.

ELIGIBILITY:
Cases Inclusion Criteria:

• Adult patients ≥18 years of age undergoing invasive mechanical ventilation in the ICU for any reason within 36 hours of intubation

Control condition A Inclusion Criteria:

• Non-invasively ventilated patients in the ICU within 36 hours of initiating non-invasive ventilation

Control condition B Inclusion Criteria

• Non-ventilated patients admitted to the ICU receiving no respiratory support or oxygen therapy alone, including high flow nasal cannula

Exclusion Criteria:

* Patients expected to be extubated within 24 hours of screening for eligibility
* Patients who have already undergone a SBT at time of screening
* Patients with a previously diagnosed neuromuscular disorder
* Patients receiving long-term invasive mechanical ventilation (prior to current hospitalization)
* Patients who have required previously (during current hospitalization) a period of invasive ventilation in ICU of more than 24 hours
* Patients who have previously been enrolled in the study
* Patients for whom post-hospital follow-up may be challenging, e.g. those who reside overseas or who have no fixed address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled in the Medical-Surgical ICU at Toronto General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life at home | Day 180
  5-level EQ-5D (EQ-5D-5L) score - The EQ-5D-5L is a validated self-reported instrument assessing quality of life at the moment questionnaire is completed. Each question is scored from 1 (no problems) to 5 (inability to perform activity) and are independently assessed.
Quality of life at home | Day 180
  Montreal Cognitive Assessment (MOCA) score - MoCA is a clinician-reported measure to assess for cognitive impairments. MoCA is scored out of 30 with scores <26 indicating cognitive impairment.

SECONDARY OUTCOMES:
Duration of ventilation | Until hospital discharge (up to 6 months)
Muscle research council score | Until day 14
  Muscle research council score, is a validated measure of muscle strength. Possible scores range from 0 (complete paralysis) to 60 (normal strength). Assessments will be made at first spontaneous breathing trial & at day 14.
Airway occlusion pressure (P0.1) | First spontaneous breathing trial (within 5 minutes of onset)
  P0.1 will be assessed during spontaneous breathing trial. Spontaneous breathing trials (SBT) are standard of care to assess if patients are able to be extubated from mechanical ventilation. A specific time frame cannot be provided as SBT are only conducted when care team deem the patient as capable.
Expiratory occlusion pressure (Pocc) | First spontaneous breathing trial (within 5 minutes of onset)
  Pocc will be assessed during spontaneous breathing trial. Spontaneous breathing trials (SBT) are standard of care to assess if patients are able to be extubated from mechanical ventilation. A specific time frame cannot be provided as SBT are only conducted when care team deem the patient as capable.
Maximal inspiratory pressure (MIP) | First spontaneous breathing trial within 30 minutes of onset
  MIP will be assessed during spontaneous breathing trial. Spontaneous breathing trials (SBT) are standard of care to assess if patients are able to be extubated from mechanical ventilation. A specific time frame cannot be provided as SBT are only conducted when care team deem the patient as capable.
Days alive and at home at 180 days post ICU discharge | Day 180
Changes in abdominal muscle thickening fraction during cough | At first spontaneous breathing trial within 30 minutes of onset and at ICU discharge, an average of 7 days
  Abdominal muscle thickening fraction during cough will be assessed by ultrasound during SBT when care team deems patient capable and safe to do so, as such a specific time frame for SBT cannot be provided. Additionally abdominal muscle thickening fraction will be assessed at ICU discharge. A specific time frame cannot be provided as ICU discharge will vary between patients.
Maximal diaphragm thickening fraction | At first spontaneous breathing trial within 30 minutes of onset and at ICU discharge, an average of 7 days
  Maximal diaphragm thickening fraction will be assessed by ultrasound during SBT when care team deems patient capable and safe to do so, as such a specific time frame for SBT cannot be provided. Additionally abdominal muscle thickening fraction will be assessed at ICU discharge. A specific time frame cannot be provided as ICU discharge will vary between patients.
Changes in resting abdominal muscle thickening | Until Day 14
  Diaphragm ultrasound to measure thickening of abdominal muscles during resting tidal breathing.
Changes in resting thickening fraction | Until Day 14
  Diaphragm ultrasound to measure thickening fraction during resting tidal breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No